CLINICAL TRIAL: NCT04164303
Title: Conservative Management of DeQuervain's Tendinopathy With an Orthopaedic Manual Therapy Approach Emphasizing First CMC Manipulation: A Retrospective Case Series
Status: Completed | Type: Observational
Sponsor: Regis University (Other)
Responsible Party: Sponsor
Other Study IDs: 1407911-2
Record Dates: First submitted 2019-06-18; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: DeQuervain's Tendinopathy
Keywords: DeQuervain's tendinopathy; CMC manipulation; Physical Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical Therapist management — Physical Therapist management included joint manipulation, mobilization with movement, strengthening exercises, and grip proprioception training.

SUMMARY:
This is a retrospective review of three patients with DeQuervain's Tendinopathy (DQT) that had successful outcomes with a manual therapy focused approach provided by Physical Therapist management.

DETAILED DESCRIPTION:
DeQuervain's tendinopathy (DQT) is a musculoskeletal disorder that limits hand function of affected individuals. Management of DQT can include splinting, activity modification, medications, corticosteroid injections, Physical Therapy, and surgery. There is limited evidence to support the combination of manual therapy and exercise interventions within an Orthopaedic Manual Physical Therapy (OMPT) approach when managing patients with DQT. Three patients identified with DQT underwent a multi-modal treatment regimen including carpometacarpal (CMC) thrust and non-thrust manipulation, end range radiocarpal mobilization, mobilization with movement (MWM), strengthening exercises, and grip proprioception training. Outcomes were assessed using the numeric pain rating scale (NPRS), Jamar hand dynamometer grip strength, and the Quick Disabilities of the Arm, Shoulder, and Hand (Quick DASH) questionnaire. These measures were administered at baseline and discharge.

ELIGIBILITY:
Inclusion Criteria:

Five or more items present on the DQT screening tool devised by Batteson et al.:

* Pain over the radial styloid
* Tenderness over the dorsal thumb
* Pain with active thumb flexion
* Localized swelling over the thumb
* Positive Finkelsteins test
* Thickening of the tendon sheath of the first dorsal extensor compartment
* Pain with resisted thumb extension.

Exclusion Criteria:

* Cardiovascular disorders
* Non-musculoskeletal complaints
* Auto-immune disorders
* Patients who had received previous treatment for their condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with DeQuervain's tendinopathy.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quick Disabilities of the Arm, Shoulder, and Hand questionnaire at 8 weeks | up to 8 weeks
  Quick DASH (0% disability to 100% disability)
Change from Baseline Numeric Pain Rating Scale at 8 weeks | up to 8 weeks
  Numeric Pain Rating Scale (0-10 point scale)
Change from Baseline Grip strength at 8 weeks | up to 8 weeks
  Jamar hand dynamometer Grip strength